CLINICAL TRIAL: NCT02400775
Title: A Study to Evaluate the Effects of Azilsartan on Coronary Artery Plaque in Essential Hypertensive Patients With Stable Angina and Dyslipidemia.
Acronym: ALIVE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Azilsartan-4001; U1111-1167-9135 (Registry Identifier: WHO); JapicCTI-152834 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-03-10; First posted 2015-03-27 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Essential Hypertension With Stable Angina and Dyslipidemia
Keywords: Pharmacotherapy
MeSH Terms: conditions — Dyslipidemias | interventions — azilsartan

ARMS (1):
- Azilsartan (Experimental): Azilsartan orally once daily in the morning, either before or after breakfast
  Interventions: Drug: Azilsartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan tablets
  Other Names: Azilva tablets

SUMMARY:
The purpose of this study is to evaluate the effects of oral azilsartan once daily for 32 weeks on coronary artery plaque in essential hypertensive patients with stable angina and dyslipidemia.

DETAILED DESCRIPTION:
The open-label design without a control group was selected because this clinical study primarily aims to explore the effects of azilsartan on coronary artery plaques.

This study targeting patients with coronary artery plaque has been designed to enroll hypertensive patients with dyslipidemia. Also in light of the invasive nature of the major assessment procedures (i.e., IB-IVUS, OCT), this study will only enroll patients with stable angina planned to undergo percutaneous coronary intervention with stent placement, among patients with coronary artery plaque.

The starting dose of azilsartan has been set to 20 mg on the basis of the usual clinical dose of the drug in patients with essential hypertension, and dose increase of azilsartan will be permitted only when the target blood pressure has not been achieved.

The duration of treatment has been set to 32 weeks in line with clinical practice, in which coronary angiography is typically performed after a 32-week follow-up period following PCI with stent placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension with office blood pressure before the start of study treatment (Week 0) meeting the following criteria who are appropriate for azilsartan therapy in the opinion of the principal investigator or investigator

   * Patients aged ≥ 75 years at the time of informed consent: Sitting systolic blood pressure ≥ 150 mmHg or sitting diastolic blood pressure ≥ 90 mmHg
   * Patients aged < 75 years at the time of informed consent who concurrently have type 2 diabetes mellitus: Sitting systolic blood pressure ≥ 130 mmHg or sitting diastolic blood pressure ≥ 80 mmHg
   * Patients aged < 75 years at the time of informed consent who concurrently have chronic kidney disease (CKD) with proteinuria: Sitting systolic blood pressure ≥ 130 mmHg or sitting diastolic blood pressure ≥ 80 mmHg
   * Patients meeting none of the above: Sitting systolic blood pressure ≥ 140 mmHg or sitting diastolic blood pressure ≥ 90 mmHg
2. Patients with stable angina with a coronary stenosis confirmed by coronary angiography who are planned to undergo percutaneous coronary intervention with stent placement (any type of stent)
3. Patients with findings of integrated backscatter intravascular ultrasound (IB-IVUS) to be performed before the start of study treatment (Week 0) showing plaque at (≥ 5 mm in length) ≥ 5 mm proximal to the proximal end of the inserted stent in the coronary artery
4. Patients with dyslipidemia meeting both of the following criteria:

   * Patients treated with one HMG-CoA reductase inhibitor with no change in the dosage for at least 12 weeks before informed consent
   * Patients with an LDL-C level of < 100 mg/dL as shown by a laboratory test performed within 4 weeks before informed consent
5. Men or women aged 20 or older at the time of informed consent
6. Patients capable of making outpatient study visits throughout the observation period
7. Patients who, in the opinion of the principal investigator or investigator, are capable of understanding the contents of the clinical study and complying with the study requirements
8. Patients capable of providing written consent in person before any study procedures

Exclusion Criteria:

1. Patients with secondary hypertension or malignant hypertension
2. Patients who took any renin-angiotensin system inhibitor within 12 weeks before informed consent
3. Patients who previously underwent coronary artery bypass grafting
4. Patients with type 1 diabetes mellitus
5. Patients with insulin therapy
6. Patients with an HbA1c level (National Glycohemoglobin Standardization Program [NGSP] value) of ≥ 7.0% as shown by a laboratory test performed within 4 weeks before informed consent
7. Patients with the plaque unevaluable because of severe calcification of the coronary artery shown by IB-IVUS to be performed before the start of study treatment (Week 0)
8. Patients with a change to their antidyslipidemic medication (including a change to the dosage) within 12 weeks before informed consent
9. Patients with clinically evident renal disorder (defined as estimated glomerular filtration rate < 30 mL/min/1.73m2)
10. Patients with severe liver disorder
11. Patients with hyperkalemia (defined as serum potassium ≥ 5.5 mEq/L)
12. Patients with a history of hypersensitivity or allergy to azilsartan
13. Patients participating in any other clinical study
14. Pregnant women, women with possible pregnancy, or breastfeeding women
15. Other patients who are inappropriate for participation in this study in the opinion of the principal investigator or investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in percentage of the lipid pool in the coronary artery plaque | 32 weeks
  Change in percentage of the lipid pool in the coronary artery plaque from the start of the treatment period at the end of the treatment period (Week 32).
  Percentage of the lipid pool in the coronary artery plaque is measured by integrated backscatter intravascular ultrasound (IB-IVUS).

SECONDARY OUTCOMES:
Change in volume of the coronary artery plaque | 32 weeks
  Change in the volume of the coronary artery plaque from the start of the treatment period to the end of the treatment period.
  Change from baseline in volume of the coronary artery plaque is measured by integrated backscatter intravascular ultrasound (IB-IVUS).
Change in percentage of the fibrotic component in the coronary artery plaque | 32 weeks
  Change in percentage of the fibrotic component in the coronary artery plaque from the start of the treatment period at the end of the treatment period (Week 32).
  Percentage of the fibrotic component in the coronary artery plaque is measured by integrated backscatter intravascular ultrasound (IB-IVUS).
Change in percentage of the calcified component in the coronary artery plaque | 32 weeks
  Change in percentage of the calcified component in the coronary artery plaque from the start of the treatment period at the end of the treatment period (Week 32).
  Percentage of the calcified component in the coronary artery plaque is measured by integrated backscatter intravascular ultrasound (IB-IVUS).
Change in number of microchannels | 32 weeks
  Change from baseline in number of microchannels is measured by Optical Coherence Tomography(OCT).
Change in thickness of the fibrous cap | 32 weeks
  Change from baseline in number of microchannels is measured by Optical Coherence Tomography(OCT).

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Tokushima, Japan